CLINICAL TRIAL: NCT06413706
Title: A Randomized, Open-Label, Phase 2 Study Evaluating Abemaciclib in Combination With Temozolomide Compared to Temozolomide Monotherapy in Children and Young Adults With Newly Diagnosed High-Grade Glioma Following Radiotherapy
Brief Title: A Study Comparing Abemaciclib Plus Temozolomide to Temozolomide Monotherapy in Children and Young Adults With High-grade Glioma Following Radiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18646; I3Y-MC-JPEH (Other: Eli Lilly and Company); 2022-502269-13-00 (EU CTIS Number); U1111-1289-0405 (Other: UTN)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Glioma
Keywords: Brain tumor; Central nervous system (CNS) tumor; Spinal cord tumor; Cyclin-dependent kinase (CDK) 4/6 inhibitor
MeSH Terms: conditions — Glioma; Brain Neoplasms; Neoplasms; Spinal Cord Neoplasms | interventions — abemaciclib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abemaciclib + Temozolomide - Arm A (Experimental): Participants will receive abemaciclib administered orally in addition to temozolomide administered orally or intravenously (IV).
  Interventions: Drug: Abemaciclib; Drug: Temozolomide
- Temozolomide - Arm B (Active Comparator): Participants will receive temozolomide administered orally or IV.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib + Temozolomide - Arm A
Drug: Temozolomide — Administered orally or IV

SUMMARY:
The purpose of this study is to measure the benefit of adding abemaciclib to the chemotherapy, temozolomide, for newly diagnosed high-grade glioma following radiotherapy.

Your participation could last approximately 11 months and possibly longer depending upon how you and your tumor respond.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven high-grade glioma (HGG) as defined by 2016 World Health Organization (WHO) Classification Criteria, Grade 3-4 including:
* Anaplastic astrocytoma
* Anaplastic ganglioglioma
* Anaplastic oligodendroglioma.
* Anaplastic pleomorphic xanthoastrocytoma,
* Glioblastoma

OR as defined by the 2021 WHO Classification Criteria as molecularly characterized:

* Non-pontine diffuse midline glioma, H3 K27-altered,
* Diffuse hemispheric glioma, H3 G34-mutant
* Diffuse pediatric HGG, H3/IDH-wildtype
* Infant-type hemispheric glioma
* High-grade astrocytoma with piloid features
* High-grade pleomorphic xanthoastrocytoma
* IDH-mutant diffuse glioma with homozygous cyclin- dependent kinase inhibitor 2A/B (CDKN2A/B) deletion,
* IDH-mutant and 1p/19q co-deleted oligodendroglioma
* IDH-mutant astrocytoma with homozygous CDKN2A/B deletion
* Contraceptive use should be consistent with local regulations for participants in clinical studies.
* Radiotherapy initiated within 6 weeks (+1 week) of diagnosis and administered over 6 weeks (±1 week). Participants <3 years of age, considered not suitable for radiotherapy may be eligible.
* Minimum of 4 weeks between completion of radiation and Cycle 1 Day 1 (C1D1).
* Maximum of 8 weeks between completion of radiation and C1D1. Exceptional circumstances can be discussed with the medical monitor.
* Acute effects of prior therapies must be Grade ≤1 unless deemed clinically insignificant by the investigator.
* Adequate hematologic and organ function ≤7 days prior to C1D1
* Life expectancy of ≥8 weeks and deemed likely to complete at least 1 cycle of treatment.
* A performance score of ≥60 using:

  1. Lansky scale for participants <16 years
  2. Karnofsky scale for participants ≥16 years
* Able to swallow and/or have a gastric/nasogastric tube.
* Any current systemic steroid use dose must be stable or decreasing at least 7 days prior to C1D1.
* Able and willing to adhere to study procedures, including frequent blood draws and MRI.
* At least 28 days since any major surgery, laparoscopic procedure, or a significant traumatic injury.
* Has a body surface area (BSA) of ≥0.2 m2.

Exclusion Criteria:

Participants are excluded if any of the following apply:

* Diffuse Intrinsic Pontine Glioma (DIPG) or diffuse midline glioma located in the pons.
* Recurrent or refractory HGG including any recurrence/progression during/after radiotherapy.
* Secondary HGG, defined as a previously treated low-grade glioma that now meets high- grade criteria, or that resulted from a previously treated malignancy.
* Have known pathogenic somatic mutations appropriate for an anaplastic lymphoma kinase (ALK), B-rapidly accelerated fibrosarcoma (BRAF), or neurotrophic tyrosine receptor kinase (NTRK ) inhibitor, in regions where these therapies are available and deemed appropriate by the investigator.
* Prior HGG treatment (including bevacizumab), except for surgery and radiotherapy (with or without concomitant temozolomide).
* Current enrollment in another trial deemed incompatible with this study.
* Treatment with an investigational product within the last 30 days or 5 half-lives (whichever is longer).
* Prior malignancy within the previous 3 years that, per the investigator and the medical monitor, may affect interpretation of study results.
* A preexisting medical condition(s) that, per the investigator, would preclude study participation.
* Any serious, active, systemic infection requiring IV antibiotic, antifungal, or antiviral therapy, including acute hepatitis B or C, or Human Immunodeficiency Virus at C1D1.
* Intolerability or hypersensitivity such as urticaria, anaphylaxis, toxic necrolysis, and/or Stevens-Johnson syndrome to temozolomide, and/or abemaciclib, their excipients, or dacarbazine.
* Received a live virus vaccine within 28 days of C1D1.
* Pregnant, breastfeeding, or intend to become pregnant during the study.

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival as Determined by Blinded Independent Review Committee | Baseline up to approximately 11 months
  Event free survival as determined by blinded independent review committee.

SECONDARY OUTCOMES:
Event Free Survival as Determined by Investigator Assessment | Baseline up to approximately 11 months
  Event free survival as determined by investigator assessment
Overall Survival (OS) | Baseline to date of death due to any cause (up to approximately 18 months)
  Overall survival
Overall Response Rate (ORR) | Baseline up to approximately 3 months
  Overall response rate
Disease Control Rate (DCR) | Baseline through to disease progression (up to approximately 3 months )
  Disease control rate
Duration of Response (DoR) | Date of Complete Response (CR) or Partial Response (PR) or Minor Response (MR) to date of disease progression or death (up to approximately 3 months )
  Duration of response
Pharmacokinetic (PK): Abemaciclib Plasma Concentration | Cycle 1 through Cycle 4 (21 Day cycle)
  PK Abemaciclib Plasma Concentrations
Abemaciclib Acceptability and Palatability Questionnaire | Day 1 of Cycles 1 through 3 (21 Day Cycles)]
  Participants evaluated abemaciclib acceptability (palatability and ease of administration) using a 5-category questionnaire. Participants were asked to select one of the following to describe the acceptability of abemaciclib: Very difficult, difficult, neither easy nor difficult, easy, or very easy.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (63):
- United States (21):
  - University of Alabama at Birmingham (UAB) - Children's Hospital - The Alabama Center for Childhood Cancer and Blood -T, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University Of California - San Diego Moores Cancer Center, La Jolla, California
  - Children's Hospital of Orange County - Orange, Orange, California
  - Lucile Packard Children's Hospital (LPCH) - Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - The University of Chicago Medicine, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - The Johns Hopkins Hospital (JHH) - Johns Hopkins Childrens Center, Baltimore, Maryland
  - University of Michigan Health System (UMHS) - C.S. Mott Children's Hospital - Hematology Oncology Clinic, Ann Arbor, Michigan
  - Corewell Health, Helen DeVos Childrens Hospital Hematology and Oncology, Grand Rapids, Michigan
  - University of Minnesota / Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University (OHSU) - Doernbecher Children's Hospital, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - UT Southwestern Medical Center Dallas/Childrens Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Australia (3):
  - Queensland Government- Lady Cilento Children's Hospital, Brisbane
  - Perth Children's Hospital, Nedlands
  - The Children's Hospital at Westmead, Westmead
- Belgium (4):
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Regional CHR de la Citadelle, Liège
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Copenhagen University Hospital-Rigshospitalet University Hospital, Copenhagen, Denmark
- France (8):
  - Centre Hospitalier Universitaire d'Angers (CHU Angers), Angers
  - Centre Hospitalier Universitaire de Bordeaux Groupe Hospitalier Pellegrin Hopital des Enfants, Bordeaux
  - Centre de Lutte Contre le Cancer (CLCC) - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital La Timone, Marseille
  - Institut Curie, Paris
  - CHU de Nancy Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy-Gustave Roussy Cancer Center -DITEP, Villejuif
- Italy (10):
  - IRCCS - AOU di Bologna - Sant¿Orsola Malpighi, Bologna
  - Instituto Giannina Gaslini, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Di Rilievo Nazionale Santobono Pausilipon, Naples
  - Instituto Oncologico Veneto, Padua
  - Universita Di Padova, Padua
  - IRCCS Ospedale Pediatrico Bambino Gesu, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - A.O.U. Citta della Salute e della Scienza di Torino - Ospedale Infantile Regina Margherita, Torino
- Japan (3):
  - Nagoya University Hospital, Nagoya
  - Osaka City General Hospital, Osaka
  - National Center for Child Health and Development (NCCHD), Setagaya-Ku Tokyo
- Princess Maxima Center for Voor Kinderoncologie B.V, Utrecht, Netherlands
- Romania (2):
  - Institutul Oncologic Prof. Dr. Alexandru Trestioreanu Bucuresti (IOB), Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca
- Spain (10):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Sant Joan de Deu Barcelona, Esplugues de Llobregat
  - Hospital Infantil Universitario Nino Jesus (HIUNJS), Madrid
  - Hospital Universitario La Paz, Madrid
  - START Madrid CIOCC Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/